CLINICAL TRIAL: NCT06556004
Title: Phase 1 Clinical Trial to Determine the Safety of TRIMELVax for Stage IIIC and IV Melanoma Patients in Progression to Immunotherapy Treatment (Checkpoint Inhibitors)
Brief Title: Phase 1 Study Using TRIMELVax for Stage IIIC / IV Melanoma Patients
Acronym: Trimelvax001
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Chile (Other)
Collaborators: Hospital del Salvador (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCHIT19I0061; IT19I0061 (Other Grant/Funding Number: FONDEF, ANID)
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2023-10

CONDITIONS: Melanoma Stage IIIc; Melanoma Stage IV
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: In this trial, 20 patients will be enrolled and treated with TRIMELVax (subcutaneous). The patients will be recruited from a hospital in the Metropolitan Region: The oncology section of Hospital del Salvador. This center currently treats patients diagnosed with unresectable or metastatic melanoma with checkpoint inhibitors immunotherapy (mainly with Nivolumab).
  If a patient withdraws consent to participate in the study (including the use of data and samples already collected) or does not start treatment due to absence or death, he or she will be replaced by another participant until the number of 20 treated participants is completed.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stage IIIC and IV melanoma patients (Experimental): TRIMELVax will be administered from 10x106 melanoma cells / mL. The dose schedule considers 4 immunizations distributed as follows: the first dose on day 0, the second dose on day 28, the third dose on day 56, and the fourth dose on day 84. Conditioned tumor lysate from 10x106 melanoma cells / mL will be administered s.c. at 500 µL / dose.
  Interventions: Biological: TRIMELVAX

INTERVENTIONS:
Biological: TRIMELVAX — The safety of this immunotherapeutic compound will be tested in patients with advanced melanoma and will secondarily evaluate the induced immune response.

SUMMARY:
A new cancer vaccine called TRIMELVax will be tested as a potential treatment for patients with unresectable stage III or stage IV melanoma who have progressed to anti-PD1 immune checkpoint blockers treatment or who have presented unacceptable toxicity to the treatment. This vaccine breaks the body's tolerance to cancer cells and triggers a specific immune response against tumors. It is made from heat-treated melanoma tumor cells combined with a natural booster. In tests with mice, the vaccine caused tumor shrinkage and activated a strong immune response against melanoma and colorectal cancer.

TRIMELVax consists of three types of human melanoma-destroyed cells that are heat-treated and mixed with a booster derived from a mollusk hemocyanin. Patients will receive four injections of the vaccine in one treatment cycle.

A Phase I clinical trial will be conducted to test the safety of TRIMELVax for stage IIIC and IV melanoma patients with unresectable stage III or stage IV melanoma who have progressed to anti-PD1 immune checkpoint blockers treatment or who have presented unacceptable toxicity to the treatment. The study includes 20 patients meeting specific criteria, such as being over 18 years old, having confirmed stage IIIC or IV melanoma, and having a good performance status.

The study's main goals are to assess potential side effects and measure the vaccine's impact on the patient's immune system. Blood samples will be taken before each treatment and monthly for the first year of follow-up. We will look for specific markers on certain immune cells to evaluate the vaccine's effectiveness. We will also conduct a test to evaluate the immune response one month after the last vaccine dose.

The study is conducted in two Chilean medical centers, the Oncology Service at the Hospital Salvador, where patients receive their standard cancer treatment and support. Our primary focus is ensuring the vaccine's safety and understanding its impact on the immune system.

DETAILED DESCRIPTION:
Cancer vaccines emerge as a promising treatment alternative for patients refractory to immune checkpoint blockers (ICBs) because vaccination can break the tolerance, generating new specific immune responses capable of modulating the tumor microenvironment. TRIMELVax is a new immunogenic formulation prototype developed for treating solid tumors. It is obtained from heat-conditioned melanoma tumor cell lysates combined with a natural adjuvant. Preclinical studies showed tumor regression in murine models challenged with melanoma and colorectal cancer, activating a robust immune response against these tumors. The present vaccine is based on three allogeneic melanoma cell lysates pre-activated by a heat shock, which includes the direct subcutaneous injection as a vaccine, combined with an adjuvant derived from a mollusk hemocyanin, in one cycle of four injections. The present phase I clinical study entitled "Phase 1 Clinical Trial to Determine the Safety of TRIMELVax for Stage IIIC and IV Melanoma Patients, in Progression to Immunotherapy Treatment (Checkpoint Inhibitors)" will include 20 stage IV melanoma patients according to the following inclusion criteria: People over 18 years old with histological confirmation of AJCC malignant melanoma Stage IIIC or IV. Performance Status 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale. Life expectancy over 3 months. Disease progression after anti-PD1 immune checkpoint blockers treatment or who have presented unacceptable toxicity to the treatment. Patients will be recruited in the Hospital del Salvador Oncology Service, where they will receive their experimental treatment and standard cancer care support.

Primary Objectives: Possible adverse effects should be evaluated to ensure the safety of the treatment and follow the CTCAE criteria (Common Terminology Criteria for Adverse Events) version 5.0. Due to the many adverse events that will be monitored, the CTCAE criteria are listed at the end of the trial protocol.

To evaluate the induction of a specific systemic immune response, peripheral blood will be drawn from the patients before each treatment administration and monthly during the first year of follow-up. Different surface and intracellular markers will be measured on CD8+ and CD4+ T lymphocytes. This group of markers was named the "rescue score," and it follows the proposal of Huang et al. (2017) and Sarhan et al. (2017) to evaluate immune responses to immunotherapies in humans. In addition, the Delayed Hypersensitivity or DTH test will be used thirty days after the last immunization to evaluate the in vivo immune response as described in López et al. (2009).

ELIGIBILITY:
Inclusion Criteria:

* People over 18 years old
* Histological confirmation of AJCC malignant melanoma Stage IIIC or IV.
* Performance Status 0 or 1 in the scale of Eastern Cooperative Oncology Group (ECOG).
* Life expectancy over 3 months
* Prior to the beginning of the study, participants should be aware of the risk information and express their willingness to participate by a written consent.
* Disease progression after the use of checkpoint inhibitors immunotherapy.

Exclusion Criteria:

* History of other cancers diagnosed in a period of less than 5 years, except for squamous or basal cell skin cancer, cervical cancer in situ or superficial bladder cancer, properly treated and cured.
* Ocular melanoma.
* Old or recent story of autoimmune disease.
* Systemic use of corticosteroids or immunosuppressants within 28 days prior to the start of the study. The use of inhalation corticosteroids is allowed.
* Adrenal insufficiency, requiring the use of corticosteroids, at any dose.
* Presence of symptomatic cardiac arrythmias, atrial fibrillation or prolongation of the QT-interval.
* Arterial hypertension that is not under control (systolic pressure higher than 160 mmHg and or diastolic pressure higher than 100 mmHg.
* History of symptomatic cardiovascular diseases over the last 12 months (unstable coronary disease, symptomatic vascular disease, heart failure/ functional capacity III or IV according to the New York Heart Association, history of cerebrovascular accident including transient ischemic attack, untreated deep vein thrombosis, pulmonary embolism).
* History of HIV, HBV and / or HCV infections
* Major surgery over the last 28 days
* History of splenectomy
* Uncontrolled infection or any known medical condition, that according to the investigator's interpretation may increase the risk involved in the participation of the study, or interfere with treatment or follow ups, or interfere with the interpretation of safety results.
* Inability to carry out the informed consent process.
* History of allogeneic bone marrow transplant.
* Ongoing pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-02 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Safety of treatment | 1 year
  The main objective is the safety of the therapy that will be evaluated in medical controls by a medical oncologist. Adverse events will be measured according to CTCAE 5.0.
  The CTAE criteria is a descriptive terminology most used in the world to report adverse events in trial therapies and that determines a severity scale for each reported adverse event. These criteria define an adverse event as any involuntary and unfavorable sign, symptom, or illness temporarily associated with the use of this therapy or procedure and that may or may not be related to it.

SECONDARY OUTCOMES:
Specific immune response | 1 year
  To evaluate the induction of a specific systemic immune response, peripheral blood will be drawn from the patients before each treatment administration and monthly during the first year of follow-up. Different surface and intracellular markers will be measured on CD8+ and CD4+ T lymphocytes. This group of markers was named the "rescue score," and it follows the proposal of Huang et al. (2017) and Sarhan et al. (2017) to evaluate immune responses to immunotherapies in humans. In addition, the Delayed Hypersensitivity or DTH test will be used thirty days after the last immunization to evaluate the in vivo immune response as described in López et al. (2009).
Objective tumor response | 1 year
  Tumor response will be measured by PET CT or CT of the thorax, abdomen, and pelvis, using the RECIST 1.1 criteria to evaluate the best response. There will be a baseline image (maximum one month prior to the start of the protocol), another at the end of the four administrations, and then every three months or until progression.
  The clinical response will also be evaluated in lesions visible on physical examination, and their progression will be sufficient to classify the patient as having progressive disease.
Progression-free survival (PFS) and overall survival (OS) | 2 years
  PFS It will be measured from the date the first cycle was administered until progression, whether evidenced by physical examination or images. OS It will be measured from the date that the first cycle was administered until the patient's death.

CONTACTS AND LOCATIONS:
Overall Officials: Flavio Salazar, PhD, Study Chair — University of Chile
Locations (2):
- Chile (2):
  - Hospital Salvador, Santiago, RM
  - Faculty of Medicine, University of Chile, Santiago, RM

IPD SHARING:
Plan to Share IPD: Yes
Anonymized protocol data will be shared upon request by other researchers via the researchers' email addresses. Applicants will be asked to provide information about their request. Information to review the results will be shared; information to carry out other studies must be reviewed by the ethics committee before delivery. A research team meeting with the applicants will be considered for an adequate response to the requests.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The data will be shared when requested by other researchers, starting in 2025, for two years.
Access Criteria: Requests to check published results with original data. Requests to perform other analyses before approval of the ethics committee. A meeting with the applicants will be considered to clarify the information.

REFERENCES:
- See also: Common Terminology Criteria for Adverse Events (CTCAE) — https://ctep.cancer.gov/protocolDevelopment/electronic_applications/ctc.htm